CLINICAL TRIAL: NCT02918344
Title: Prospective Study: Complications From the Use of Calcium Phosphate Paste in Mandibular Lengthening Osteotomies
Brief Title: Complications From the Use of Calcium Phosphate Paste in Mandibular Lengthening Osteotomies
Status: Completed | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: Calciumfosfaat cement
Record Dates: First submitted 2016-09-27; First posted 2016-09-28 (Estimated); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Jaw Anomalies; Infection
Keywords: calcium phosphate paste
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — microbiological smear in case of infection
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Standard sagittal split osteotomy group: Patients undergoing sagittal split osteotomy without paste application
  Interventions: Other: Hydroset; Procedure: Standard sagittal split osteotomy
- Cohort/Hydroset group: Patients undergoing sagittal split osteotomy with paste application
  Interventions: Other: Hydroset; Procedure: Standard sagittal split osteotomy

INTERVENTIONS:
Other: Hydroset — Calcium phosphate paste is used in mandibular lengthening surgery to avoid an unaesthetic notching at the lower border and to help stabilize the segments when osteosynthesis slippage is feared for.
Procedure: Standard sagittal split osteotomy — The sagittal split osteotomy (SSO) is commonly used to correct dentofacial discrepancies.

SUMMARY:
The goal of this study is to determine if the use of calcium phosphate paste in mandibular lengthening surgery causes more complications as surgical site infections and hardware removal.

An evaluation will be made to determine if the benefits of the use of the paste (3D-stability, prevention of early relapse and unaesthetic indentation) outweighs the disadvantages.

DETAILED DESCRIPTION:
The sagittal split osteotomy (SSO) is commonly used to correct dentofacial discrepancies. Correction of distocclusion can be achieved through lengthening of the mandible, and a balanced facial appearance can be obtained by increasing chin projection.

Calcium phosphate paste is used in mandibular lengthening surgery to avoid an unaesthetic notching at the lower border(1)(2) and to help stabilize the segments when osteosynthesis slippage is feared for. A recently performed retrospective study showed an increase of infectious complications when calcium phosphate paste was used for this indications. Several precautions were identified that could be undertaken to decrease the infectious complications. The study concluded that a prospective study was required in which these precautions were implemented to determine whether infectious complications can be reduced.

The aim of this study is to investigate whether the hardened paste still increases the incidence of site infections after implementation of several precautions and the use of a standardized antibiotic prophylactic protocol.

ELIGIBILITY:
Inclusion Criteria:

* All patients with dysgnatic deformities requiring mandibular lengthening surgery
* Gender: M/F
* Age: >15y-75y

Exclusion Criteria:

* Previous orthognathic surgery
* Congenital facial malformations
* Unilateral SSO
* Immunodeficiency
* Simultaneous removal of lower third molars
* Incomplete postoperative follow-up

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing bilateral sagittal split osteotomy
Sampling Method: Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Surgical site infection | 6 months
  Determine the number of surgical site infection

SECONDARY OUTCOMES:
Hardware removal | 6 months
  Determine the number of hardware removal
Revision | 6 months
  Determine the number of revisions

CONTACTS AND LOCATIONS:
Overall Officials: Erica Coppey, Dr., Principal Investigator — Universitair Ziekenhuis Brussel; Maurice Mommaerts, Prof.Dr.Mult, Study Director — Universitair Ziekenhuis Brussel
Locations (1):
- universitair Ziekenhuis brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No